CLINICAL TRIAL: NCT04415801
Title: Effect of Repeated Removal and Re-placement of Laser Microgrooved and Machined Abutments on Proinflammatory Cytokine Levels Around Dental Implants
Brief Title: Effect of Repeated Removal and Re-placement of Abutments Around Dental Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Renzo Guarnieri, Adjunct Professor, University of Roma La Sapienza
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 3/20
Record Dates: First submitted 2020-05-24; First posted 2020-06-04 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Peri-implant Mucositis
Keywords: Peri-implant Mucositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implant abutments (Experimental): implant abutments
  Interventions: Diagnostic Test: Repeated removal and re-placement of healing and prosthetic abutments

INTERVENTIONS:
Diagnostic Test: Repeated removal and re-placement of healing and prosthetic abutments — Repeated removal and re-placement of healing and prosthetic abutments

SUMMARY:
Repeated removal and re-placement of healing and prosthetic abutments result in frequent injuries to the soft tissues. The purpose was to evaluate the effect of repeated removal and re-placement of laser microgrooved and smooth/machined healing and prosthetic abutments during restorative stages, and 1 year after functional loading, on proinflammatory cytokine levels around dental implants.

DETAILED DESCRIPTION:
Twenty-four patients each received 2 one-stage implants in a split mouth design on the same jaw. In each patient one healing and prosthetic abutments with a laser microgrooved surface (LMS group) and one healing and prosthetic abutments with smooth/machined surface (S/MS group) were used. Four months following implant placement [Baseline (BSL)], the healing abutments were disconnnected and reconnected three times to carry out the impression procedures and metal framework try-in. Four weeks later (T0), definitive prosthetic abutments were installated with screw retained crowns. Samples for immunological analyses were taken from the sulcus around each implant at BSL, T0, and 1 year after functional loading (T1). Peri-implant crevicular fluid samples were analyzed for interleukin-1beta (IL-1β), interleukin-6 (IL-6) and tumor necrosis factor (TNF)-α levels using the ELISA kit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, in good general health, and with sufficient amount of bone available to place a standard implant

Exclusion Criteria:

* natural teeth adjacent to surgical area affected by untreated periodontal or endodontic infections, peri-implant bone defects requiring bone augmentation, absence of opposing occlusion,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline to 8 weeks of gingival fluid production | 8 weeks
  The gingival fluid production was measured electronically in Periotron units, (Periotron 8000®, Ora Flow, Inc., Plainview, NY, USA) which were converted to microliters (μl) by MCCONVRT software (Ora Flow).

CONTACTS AND LOCATIONS:
Overall Officials: Renzo Guarnieri, Principal Investigator — University La Sapienza Roma Italy
Locations (1):
- Universita la Sapienza, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guarnieri R, Miccoli G, Reda R, Mazzoni A, Di Nardo D, Testarelli L. Laser microgrooved vs. machined healing abutment disconnection/reconnection: a comparative clinical, radiographical and biochemical study with split-mouth design. Int J Implant Dent. 2021 Mar 17;7(1):19. doi: 10.1186/s40729-021-00301-6. PMID 33728493